CLINICAL TRIAL: NCT01852071
Title: Autologous Transplantation of Bone Marrow CD34+ Stem/Progenitor Cells After Addition of a Normal Human ADA Complementary DNA (cDNA) by the EFS-ADA Lentiviral Vector for Severe Combined Immunodeficiency Due to Adenosine Deaminase Deficiency (ADA-SCID)
Brief Title: Autologous CD34+ Hematopoietic Stem Cells Transduced ex Vivo With Elongation Factor 1 Alpha Shortened (EFS) Lentiviral Vector Encoding for the Human ADA Gene
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Human Genome Research Institute (NHGRI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Orchard Therapeutics (Industry)
Responsible Party: Principal Investigator, Donald B. Kohn, M.D., Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFS-ADA; U01AI100801 (NIH); 2P01HL073104 (NIH); 0910-1006 (Other: OBA-RAC)
Record Dates: First submitted 2013-05-07; First posted 2013-05-13 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: ADA-SCID
Keywords: gene therapy; hematopoietic stem cell; ADA-SCID; lentiviral vector
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Gene Therapy (Experimental): Infusion of autologous EFS-ADA Lentiviral (LV) CD34+ cells
  Interventions: Genetic: Infusion of autologous EFS-ADA LV CD34+ (OTL-101); Drug: busulfan; Drug: PEG-ADA ERT

INTERVENTIONS:
Genetic: Infusion of autologous EFS-ADA LV CD34+ (OTL-101) — autologous EFS-ADA LV CD34+ cells (OTL-101) are infused intravenously
  Other Names: OTL-101
Drug: busulfan — Busulfan is used for non-myeloablative conditioning
Drug: PEG-ADA ERT — PEG-ADA ERT is discontinued at Day +30 (-3/+15 days) after successful engraftment

SUMMARY:
The aim of this study is to assess the safety and efficacy of autologous transplantation of hematopoietic stem cells (CD34+ cells) from the bone marrow (BM) of ADA-deficient SCID infants and children following human ADA cDNA transfer by the EFS-ADA lentiviral vector. The level of gene transfer in blood cells and immune function will be measured as endpoints.

DETAILED DESCRIPTION:
The study is open to twenty (20) infants and children diagnosed with ADA-deficient SCID who did not have a medically eligible, human leukocyte antigen (HLA)-identical sibling donor for bone marrow transplantation. The EFS-ADA lentiviral vector with the human ADA cDNA will be used to transduce autologous CD34+ cells from the bone marrow of these subjects. The subjects will receive 4 mg/kg busulfan prior to re-infusion of their gene-modified cells. Safety is the primary endpoint. During the follow-up phase, the investigators aim to determine whether the cells could engraft and produce mature cells that contain and express the corrected ADA gene in the absence of pegademase bovine (PEG-ADA) enzyme replacement therapy (ERT), which will be withheld at Day +30 following transplant. Efficacy studies to evaluate the level of immune reconstitution, will be performed in the first and second years of the study.

ELIGIBILITY:
Inclusion Criteria:

-Children ≥ 1.0 months of age with a diagnosis of ADA-deficient SCID based on A. Decreased ADA enzymatic activity in erythrocytes, leukocytes, skin fibroblasts, or in cultured fetal cells to levels consistent with ADA-deficient SCID as determined by reference laboratory or confirmed ADA gene mutation(s) known to cause disease , AND

B. Evidence of severe combined immunodeficiency based on either:

1. Family history of first order relative with ADA deficiency and clinical and laboratory evidence of severe immunologic deficiency, OR
2. Evidence of severe immunologic deficiency in subject prior to institution of immune restorative therapy, based on

   1. lymphopenia (absolute lymphocyte count <400 cells/mcL) OR absence or low number of T cells (absolute CD3+ count <300 cells/mcL) OR
   2. severely decreased T lymphocyte blastogenic responses to phytohemagglutinin (either <10% of lower limit of normal controls for the diagnostic laboratory, <10% of the response of the normal control of the day, or stimulation index <10)

      * Ineligible for matched sibling allogeneic bone marrow transplantation: absence of a medically eligible HLA-identical sibling, with normal immune function, who may serve as an allogeneic bone marrow donor
      * Signed written informed consent according to guidelines of the Institutional Review Board (IRB) (UCLA Office of Human Research Protection Program and National Human Genome Research Institute (NHGRI) IRB

Exclusion Criteria:

1. Age ≤ 1.0 months Appropriate organ function as outlined below must be observed within 60 days of entering this trial.
2. Hematologic

   1. Anemia (hemoglobin < 10.5 g/dl at < 2 years of age, or < 11.5 g/dl at > 2 years of age).
   2. Neutropenia (absolute granulocyte count <500/mm3.
   3. Thrombocytopenia (platelet count < 150,000/mm3, at any age).
   4. International Normalised Ratio (INR) or Prothrombin Time (PT) > 2 times the upper limits of normal or Partial Thromboplastin Time (PTT) > 2.33 times the upper limit of normal (patients with a correctable deficiency controlled on medication will not be excluded).
   5. Cytogenetic abnormalities on peripheral blood or bone marrow or amniotic fluid (if available).
   6. Prior allogeneic Hematopoietic Stem Cell Transplant (HSCT) with cytoreductive conditioning
3. Infectious

   a. Evidence of infection with HIV-1, hepatitis B, Hepatitis C, or parvovirus B 19 by DNA Polymerase Chain Reaction (PCR) within 90 days prior to bone marrow harvest. If other infection is present, it must be under control (e.g. stable or decreasing viral load) at the time of screening
4. Pulmonary

   1. Resting O2 saturation by pulse oximetry < 95% on room air.
   2. Chest x-ray indicating active or progressive pulmonary disease.
5. Cardiac

   1. Abnormal electrocardiogram (EKG) indicating cardiac pathology.
   2. Uncorrected congenital cardiac malformation with clinical symptomatology.
   3. Active cardiac disease, including clinical evidence of congestive heart failure, cyanosis, hypotension.
   4. Poor cardiac function as evidenced by LV ejection fraction < 40% on echocardiogram.
6. Neurologic

   1. Significant neurologic abnormality by examination.
   2. Uncontrolled seizure disorder.
7. Renal

   1. Renal insufficiency: serum creatinine >= 1.2 mg/dl, or >= 3+ proteinuria.
   2. Abnormal serum sodium, potassium, calcium, magnesium, phosphate at grade III or IV by Division of AIDS Toxicity Scale.
8. Hepatic/GI:

   1. Serum transaminases > 5 times the upper limit of normal (ULN).
   2. Serum bilirubin > 2 times ULN.
   3. Serum glucose > 1.5 times ULN.
   4. Intractable severe diarrhea.
9. Oncologic

   1. Evidence of active malignant disease other than dermatofibrosarcoma protuberans (DFSP)
   2. Evidence of DFSP expected to require anti-neoplastic therapy within the 5 years following the infusion of genetically corrected cells
   3. Evidence of DFSP expected to be life limiting within the 5 years following the infusion of genetically corrected cells
10. Known sensitivity to Busulfan
11. General

    1. Expected survival < 6 months.
    2. Pregnant.
    3. Major congenital anomaly.
    4. Ineligible for autologous HSCT by the criteria at the clinical site.
    5. Other conditions which in the opinion of the principal investigator and/or co-investigators, contra-indicate the bone marrow harvest, the administration of busulfan, infusion of transduced cells or indicate the patient or patient's parents/primary caregivers inability to follow protocol.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2013-08-02 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald B Kohn, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Mattel Children's Hospital, UCLA, Los Angeles, California
  - Mark O. Hatfield Clinical Research Center, NIH, Bethesda, Maryland

REFERENCES:
- [Background] Candotti F, Shaw KL, Muul L, Carbonaro D, Sokolic R, Choi C, Schurman SH, Garabedian E, Kesserwan C, Jagadeesh GJ, Fu PY, Gschweng E, Cooper A, Tisdale JF, Weinberg KI, Crooks GM, Kapoor N, Shah A, Abdel-Azim H, Yu XJ, Smogorzewska M, Wayne AS, Rosenblatt HM, Davis CM, Hanson C, Rishi RG, Wang X, Gjertson D, Yang OO, Balamurugan A, Bauer G, Ireland JA, Engel BC, Podsakoff GM, Hershfield MS, Blaese RM, Parkman R, Kohn DB. Gene therapy for adenosine deaminase-deficient severe combined immune deficiency: clinical comparison of retroviral vectors and treatment plans. Blood. 2012 Nov 1;120(18):3635-46. doi: 10.1182/blood-2012-02-400937. Epub 2012 Sep 11. PMID 22968453
- [Background] Carbonaro DA, Zhang L, Jin X, Montiel-Equihua C, Geiger S, Carmo M, Cooper A, Fairbanks L, Kaufman ML, Sebire NJ, Hollis RP, Blundell MP, Senadheera S, Fu PY, Sahaghian A, Chan RY, Wang X, Cornetta K, Thrasher AJ, Kohn DB, Gaspar HB. Preclinical demonstration of lentiviral vector-mediated correction of immunological and metabolic abnormalities in models of adenosine deaminase deficiency. Mol Ther. 2014 Mar;22(3):607-622. doi: 10.1038/mt.2013.265. Epub 2013 Nov 20. PMID 24256635
- [Derived] Kohn DB, Booth C, Shaw KL, Xu-Bayford J, Garabedian E, Trevisan V, Carbonaro-Sarracino DA, Soni K, Terrazas D, Snell K, Ikeda A, Leon-Rico D, Moore TB, Buckland KF, Shah AJ, Gilmour KC, De Oliveira S, Rivat C, Crooks GM, Izotova N, Tse J, Adams S, Shupien S, Ricketts H, Davila A, Uzowuru C, Icreverzi A, Barman P, Campo Fernandez B, Hollis RP, Coronel M, Yu A, Chun KM, Casas CE, Zhang R, Arduini S, Lynn F, Kudari M, Spezzi A, Zahn M, Heimke R, Labik I, Parrott R, Buckley RH, Reeves L, Cornetta K, Sokolic R, Hershfield M, Schmidt M, Candotti F, Malech HL, Thrasher AJ, Gaspar HB. Autologous Ex Vivo Lentiviral Gene Therapy for Adenosine Deaminase Deficiency. N Engl J Med. 2021 May 27;384(21):2002-2013. doi: 10.1056/NEJMoa2027675. Epub 2021 May 11. PMID 33974366

RESULTS

PARTICIPANT FLOW:
Groups:
- Gene Therapy: Infusion of autologous CD34+ cells genetically modified by the EF1αS-ADA (EFS-ADA) lentiviral vector (LV)
  Busulfan: Busulfan is used for non-myeloablative conditioning
  Polyethylene glycol-modified adenosine deaminase (PEG-ADA): PEG-ADA enzyme replacement therapy (ERT) is discontinued at Day 30 +/- 3 days from date of infusion of OTL-101.
- Historical Control Group: Historical data from patients with Severe Combined Immunodeficiency Due to ADA Deficiency (ADA-SCID) who were treated with Hematopoietic Stem Cell Transplantation (HSCT): Historical data from a database of ADA-SCID patients treated with allogeneic HSCT from Great Ormond Street Hospital (GOSH) and Duke University Children's Hospital were collected as comparator group.
Period: Overall Study
Arm/Group | Gene Therapy | Historical Control Group
Started | 20 | 26
Completed | 20 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gene Therapy | Historical Control Group | Total
Number analyzed (Participants) | 20 | 26 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 26 | 46
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex, n: Female | 11 | 0 | 11
  Sex, n: Male | 9 | 0 | 9
  Sex, n: Not Reported | 0 | 26 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Hispanic | 6 | 0 | 6
  Native American or Alaska Native | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  White | 10 | 0 | 10
  Other | 3 | 0 | 3
  Unknown | 1 | 0 | 1
  Not Reported | 0 | 26 | 26
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 30
  United Kingdom | 0 | 16 | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) of Subjects Treated With Investigational Medicinal Product (IMP) (1 Year)
Description: Overall survival is defined as the percentage of subjects alive at 12 months post- treatment with OTL-101 or HSCT
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- OTL-101 Gene Therapy: The primary efficacy population consists of all subjects treated with OTL-101 at University of California, Los Angeles/National Institutes of Health (UCLA/NIH)
- HSCT Controls Without MRD: The primary comparator population from the HSCT historical control group consists of ADA-SCID patients without a medically eligible human leukocyte antigen (HLA)-identical sibling or family donor and treated with HSCT at either GOSH or Duke University between 2000 and 2016.
- HSCT Controls With MRD: ADA-SCID patients with an Matched Related Donor (MRD) treated with HSCT at either GOSH or Duke University from 2000 to 2016
- All HSCT Control Group: The complete HSCT historical control group, which consists of ADA-SCID patients with any type of donor treated with HSCT at either GOSH or Duke University from 2000 to 2016
Arm/Group | OTL-101 Gene Therapy | HSCT Controls Without MRD | HSCT Controls With MRD | All HSCT Control Group
Number analyzed (Participants) | 20 | 14 | 12 | 26
percentage of participants | 100 [83.16 to 100] | 85.71 [57.19 to 98.22] | 100 [73.54 to 100] | 92.31 [74.87 to 99.05]
Statistical Analysis 1: Comparison: OTL-101 Gene Therapy vs HSCT Controls Without MRD; Percentage of patients alive at 1-year post-treatment in the historical control groups (without MRD) were compared to the percentage of study patients alive at 1-year post-treatment with OTL-101. Results are reported as percentage difference in OS of historical control group from OTL-101 on-study subjects; Test type: Superiority; Difference in percentages = 14.29, 95% CI 2-sided [-5.40 to 42.81]
Statistical Analysis 2: Comparison: OTL-101 Gene Therapy vs HSCT Controls With MRD; Percentage of patients alive at 1-year post-treatment in the historical control groups (with MRD) were compared to the percentage of study patients alive at 1-year post-treatment with OTL-101. Results are reported as percentage difference in OS of historical control group from OTL-101 on-study subjects; Test type: Superiority; Difference in percentages = 0
Statistical Analysis 3: Comparison: OTL-101 Gene Therapy vs All HSCT Control Group; Percentage of patients alive at 1-year post-treatment in the historical control groups (all control patients) were compared to the percentage of study patients alive at 1-year post-treatment with OTL-101. Results are reported as percentage difference in OS of historical control group from OTL-101 on-study subjects; Test type: Superiority; Difference in percentages = 7.69, 95% CI 2-sided [-10.08 to 25.13]

2. Primary Outcome: Event-free Survival (EvFS) of Subjects Treated With Investigational Medicinal Product (IMP) (1 Year)
Description: Event-free survival is defined as the percentage of subjects alive with no "event", an "event" being the resumption of PEG-ADA ERT or the need for a rescue allogeneic Hematopoietic Stem Cell Transplant (HSCT), or death.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- OTL-101 Gene Therapy: The primary efficacy population consists of all subjects treated with OTL-101 at UCLA/NIH
- HSCT Controls Without MRD: The primary comparator population from the HSCT historical control group consists of ADA-SCID patients without a medically eligible HLA-identical sibling or family donor and treated with HSCT at either GOSH or Duke University between 2000 and 2016.
- HSCT Controls With MRD: ADA-SCID patients with an MRD treated with HSCT at either GOSH or Duke University from 2000 to 2016
Arm/Group | OTL-101 Gene Therapy | HSCT Controls Without MRD | HSCT Controls With MRD | All HSCT Control Group
Number analyzed (Participants) | 20 | 14 | 12 | 26
percentage of participants | 100 [83.16 to 100] | 64.29 [35.14 to 87.24] | 100 [73.54 to 100] | 80.77 [60.65 to 93.45]
Statistical Analysis 1: Comparison: OTL-101 Gene Therapy vs HSCT Controls Without MRD; Percentage of patients with EvFS at 1-year post-treatment in the historical control groups (without MRD) were compared to the percentage of study patients with EvFS at 1-year post-treatment with OTL-101. Results are reported as percentage difference in EvFS of historical control group from OTL-101 on-study subjects; Test type: Superiority; Difference in percentages = 35.71, 95% CI 2-sided [11.21 to 64.86]
Statistical Analysis 2: Comparison: OTL-101 Gene Therapy vs HSCT Controls With MRD; Percentage of patients with EvFS at 1-year post-treatment in the historical control groups (with MRD) were compared to the percentage of study patients with EvFS at 1-year post-treatment with OTL-101. Results are reported as percentage difference in EvFS of historical control group from OTL-101 on-study subjects; Test type: Superiority; Difference in percentages = 0
Statistical Analysis 3: Comparison: OTL-101 Gene Therapy vs All HSCT Control Group; Percentage of patients with EvFS at 1-year post-treatment in the historical control groups (all control patients) were compared to the percentage of study patients with EvFS at 1-year post-treatment with OTL-101. Results are reported as percentage difference in EvFS of historical control group from OTL-101 on-study subjects; Test type: Superiority; Difference in percentages = 19.23, 95% CI 2-sided [0.71 to 39.35]

3. Secondary Outcome: OS of Subjects Treated With Investigational Medicinal Product (IMP) (2 Years)
Description: OS is defined as the percentage of subjects alive at 24 months post- treatment with OTL-101 or HSCT
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OTL-101 Gene Therapy | HSCT Controls Without MRD | HSCT Controls With MRD | All HSCT Control Group
Number analyzed (Participants) | 20 | 14 | 12 | 26
percentage of participants | 100 [83.16 to 100] | 85.71 [57.19 to 98.22] | 90.91 [58.72 to 99.77] | 88.00 [68.78 to 97.45]
Statistical Analysis 1: Comparison: OTL-101 Gene Therapy vs HSCT Controls Without MRD; Percentage of patients alive at 2-years post-treatment in the historical control groups (without MRD) were compared to the percentage of study patients alive at 2-years post-treatment with OTL-101. Results are reported as percentage difference in OS of historical control group from OTL-101 on-study subjects; Test type: Superiority; Difference in percentages = 14.29, 95% CI 2-sided [-5.40 to 42.81]
Statistical Analysis 2: Comparison: OTL-101 Gene Therapy vs HSCT Controls With MRD; Percentage of patients alive at 2-years post-treatment in the historical control groups (with MRD) were compared to the percentage of study patients alive at 2-years post-treatment with OTL-101. Results are reported as percentage difference in OS of historical control group from OTL-101 on-study subjects; Test type: Superiority; Difference in percentages = 9.09, 95% CI 2-sided [-9.55 to 41.28]
Statistical Analysis 3: Comparison: OTL-101 Gene Therapy vs All HSCT Control Group; Percentage of patients alive at 2-years post-treatment in the historical control groups (all control patients) were compared to the percentage of study patients alive at 2-years post-treatment with OTL-101. Results are reported as percentage difference in OS of historical control group from OTL-101 on-study subjects; Test type: Superiority; Difference in percentages = 12.00, 95% CI 2-sided [-5.62 to 31.22]

4. Secondary Outcome: EvFS of Subjects Treated With Investigational Medicinal Product (IMP) (2 Years)
Description: Event-free survival is defined as the percentage of subjects alive with no "event", an "event" being the resumption of PEG-ADA ERT or the need for a rescue allogenic Hematopoietic Stem Cell Transplant (HSCT), or death.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OTL-101 Gene Therapy | HSCT Controls Without MRD | HSCT Controls With MRD | All HSCT Control Group
Number analyzed (Participants) | 20 | 14 | 12 | 26
percentage of participants | 100 [83.16 to 100] | 50.00 [23.04 to 76.96] | 63.64 [30.79 to 89.07] | 56.00 [34.93 to 75.60]
Statistical Analysis 1: Comparison: OTL-101 Gene Therapy vs HSCT Controls Without MRD; Percentage of patients with EvFS at 2-years post-treatment in the historical control groups (without MRD) were compared to the percentage of study patients with EvFS at 2-years post-treatment with OTL-101. Results are reported as percentage difference in EvFS of historical control group from OTL-101 on-study subjects; Test type: Superiority; Difference in percentages = 50.00, 95% CI 2-sided [22.71 to 76.96]
Statistical Analysis 2: Comparison: OTL-101 Gene Therapy vs HSCT Controls With MRD; Percentage of patients with EvFS at 2-years post-treatment in the historical control groups (with MRD) were compared to the percentage of study patients with EvFS at 2-years post-treatment with OTL-101. Results are reported as percentage difference in EvFS of historical control group from OTL-101 on-study subjects; Test type: Superiority; Difference in percentages = 36.36, 95% CI 2-sided [9.80 to 69.21]
Statistical Analysis 3: Comparison: OTL-101 Gene Therapy vs All HSCT Control Group; Percentage of patients with EvFS at 2-years post-treatment in the historical control groups (all control patients) were compared to the percentage of study patients with EvFS at 2-years post-treatment with OTL-101. Results are reported as percentage difference in EvFS of historical control group from OTL-101 on-study subjects; Test type: Superiority; Difference in percentages = 44.00, 95% CI 2-sided [22.78 to 65.23]

5. Secondary Outcome: Vector Copy Number (VCN) in Peripheral Blood (PB) Granulocytes.
Description: Vector copy number in the PB granulocyte fraction that was T cell depleted, is a surrogate for amount of engrafted genetically modified Hematopoietic stem cell (HSC) that are producing granulocytes every 3-5 days. VCN analysis was performed by Droplet Digital PCR (ddPCR) on DNA extracted from peripheral blood granulocytes.
Time Frame: 24 months
Population: Historical control groups/arms are not included in the analysis population for this outcome measure as these subjects did not receive gene therapy, and so measurement of VCN levels is not relevant
Measure: Median (Full Range); unit: copies/cell
Arm/Group | OTL-101 Gene Therapy
Number analyzed (Participants) | 18
copies/cell | 0.093 [0.04 to 2.50]

6. Secondary Outcome: VCN in Peripheral Blood Mononuclear Cells (PBMCs)
Description: PBMC VCN is a measure of the accumulation of peripheral blood leukocytes arising from engrafted, genetically modified HSC. VCN analysis was performed by ddPCR on DNA extracted from PBMC.
Time Frame: 24 months
Population: as for outcome 5
Measure: Median (Full Range); unit: copies/cell
Arm/Group | OTL-101 Gene Therapy
Number analyzed (Participants) | 18
copies/cell | 0.972 [0.13 to 1.86]

7. Secondary Outcome: ADA Activity in Erythrocytes
Description: ADA enzyme activity measured to assess the amount of functional gene product produced from the normal ADA transgene delivered by EFS-ADA LV; persistence of ADA enzyme activity over time demonstrates successful engraftment and differentiation of genetically modified HSC.
Time Frame: 24 months
Measure: Median (Full Range); unit: nmol/h/mg
Arm/Group | OTL-101 Gene Therapy | HSCT Controls Without MRD | HSCT Controls With MRD | All HSCT Control Group
Number analyzed (Participants) | 14 | 4 | 3 | 7
nmol/h/mg | 105.50 [34.1 to 268.9] | 48.500 [0.00 to 123.00] | 1.000 [1.00 to 2.00] | 2.000 [0.00 to 123.00]

8. Secondary Outcome: Reduction in Deoxyadenosine Nucleotide (dAXP) in Erythrocytes
Description: Decreased dAXP levels coincide with increased ADA enzyme activity, detoxification was used to demonstrate functional ADA enzyme production from the introduced ADA transgene. The threshold for detoxification was <100 μmol/L.
Time Frame: 24 months
Population: HSCT Controls With MRD arm is not included in the analysis population for this outcome measure as dAXP data was not reported between 17-30 months post-HSCT for any patients in this arm.
Measure: Median (Full Range); unit: umol/mL
Arm/Group | OTL-101 Gene Therapy | HSCT Controls Without MRD | All HSCT Control Group
Number analyzed (Participants) | 14 | 5 | 5
umol/mL | 0.0330 [0.007 to 0.101] | 0.0360 [0.004 to 0.256] | 0.0360 [0.004 to 0.256]

9. Secondary Outcome: Change From Baseline in CD3+ T Cell Counts (2 Years)
Description: Immune reconstitution was assessed by change in CD3+ T Cell counts at baseline to Month 24.
Time Frame: 24 months
Measure: Median (Full Range); unit: cells/μL
Arm/Group | OTL-101 Gene Therapy | HSCT Controls Without MRD | HSCT Controls With MRD | All HSCT Control Group
Number analyzed (Participants) | 14 | 5 | 1 | 6
cells/μL | 569.0 [-426 to 2211] | 340.0 [-23 to 1243] | 538.0 [538 to 538] | 395.5 [-23 to 1243]

10. Secondary Outcome: Number of Single Integration Sites Representing >30% of the Total Integration Sites (2 Years)
Description: Vector Integration Site Analysis (VISA) allowed determination of the distribution of vector integration sites in each subject's genome, as well as the relative clonal abundance. VISA was to be considered abnormal for a subject if, in 2 or more instances during the course of follow-up, a single integration site was found to represent >30% of the total integration sites detected.
Time Frame: 24 months
Population: Historical control groups/arms are not included in the analysis population for this outcome measure as these subjects did not receive gene therapy, and so measurement of VISA is not relevant
Measure: Number; unit: number of participants
Groups:
- OTL-101 Gene Therapy: The primary safety population consists of all subjects treated with OTL-101 at UCLA/NIH
Arm/Group | OTL-101 Gene Therapy
Number analyzed (Participants) | 19
number of participants | 0

11. Secondary Outcome: Severe Infection Rate Excluding the First Three Months After Treatment
Description: The infections of interest in this study were severe infections or opportunistic infectious episodes, defined as infections requiring hospitalization or prolonging hospitalization and/or documented infections by opportunistic pathogens. Infections that took place in the first 3 months of follow-up post treatment were excluded from calculations to avoid possible bias introduced in the data by the effects of conditioning.
Time Frame: 24 months
Measure: Number; unit: Infection rate per person per year
Arm/Group | OTL-101 Gene Therapy | HSCT Controls Without MRD | HSCT Controls With MRD | All HSCT Control Group
Number analyzed (Participants) | 20 | 13 | 12 | 25
Infection rate per person per year | 0.20 | 0.56 | 0.15 | 0.36

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of participant consent, approximately 1-month pre-treatment, up until 2-years post-treatment with OTL-101
Description: Adverse events were reported for subjects treated with OTL-101.
  Adverse event reporting is not applicable for the historical control arms (without MRD, with MRD, and all control patients) as this data was not collected due to the historical nature of the population.
Groups:
- OTL-101 Gene Therapy: The safety population consists of all subjects treated with OTL-101 at UCLA/NIH
Arm/Group | OTL-101 Gene Therapy
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 9/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTL-101 Gene Therapy (N=20)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (2)
Bronchiolitis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Immune reconstitution inflammatory syndrome (Immune system disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTL-101 Gene Therapy (N=20)
Neutropenia (Blood and lymphatic system disorders) | 17 (31)
Anemia (Blood and lymphatic system disorders) | 13 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (8)
Rhinovirus infection (Infections and infestations) | 4 (4)
Otitis media (Infections and infestations) | 4 (8)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Parainfluenzae virus infection (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 2 (2)
Ear infection (Infections and infestations) | 1 (2)
Aspergillus infection (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Molluscum contagiosum (Infections and infestations) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 9 (14)
Aspartate aminotransferase increased (Investigations) | 9 (11)
Transaminases increased (Investigations) | 2 (3)
Hepatic enzyme increased (Investigations) | 1 (2)
Body temperature decreased (Investigations) | 1 (1)
Epstein-Barr virus test positive (Investigations) | 1 (1)
Influenza B virus test (Investigations) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (8)
Vomiting (Gastrointestinal disorders) | 7 (14)
Constipation (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 6 (9)
Rash (Skin and subcutaneous tissue disorders) | 5 (8)
Eczema (Skin and subcutaneous tissue disorders) | 4 (5)
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 (3)
Skin lesion (Skin and subcutaneous tissue disorders) | 3 (3)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (11)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyrexia (General disorders) | 7 (9)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Ear injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Blepharospasm (Eye disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT01852071/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/71/NCT01852071/SAP_001.pdf